CLINICAL TRIAL: NCT02665078
Title: Feasibility of a Minimally Invasive Thoracoscopic Ultrasound for Localization of Pulmonary Nodules Using Resected Human Lungs
Brief Title: Feasibility of a Minimally Invasive Thoracoscopic Ultrasound for Localization of Pulmonary Nodules
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 13-7111
Record Dates: First submitted 2015-05-15; First posted 2016-01-27 (Estimated); Last update posted 2018-02-26 (Actual); Status verified 2018-02

CONDITIONS: Lung Cancer
Keywords: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Thoracoscopic Ultrasound: Patients who undergo lobectomy or an anatomical segmental resection for malignant lung tumors will be enrolled in the study. After lung resection, the lung will be evaluated by XLTF-UC180 for localization of the tumor. The ultrasound probe will be put on the lung surface in several different directions to obtain the cross section with maximum diameter. The ultrasound image with size measurement of the tumor will be recorded using an ultrasound scanner (EU-Y0008, OLYMPUS MEDICALSYSTEMS CORP., Tokyo, Japan). After ultrasound evaluation, the specimen will be delivered directory to the pathology laboratory and the actual tumor size and histological diagnosis will be determined. In addition, we will evaluate the differences between US image and pathological morphology using HE slides of lung tumor.
  Interventions: Other: Thoracoscopic Ultrasound

INTERVENTIONS:
Other: Thoracoscopic Ultrasound — We will evaluate the resected specimen using the XLTF-UC180 in the operating room (OR) to determine the localization rate of the targets. Ultrasound measurement and images will be compared to the actual size of the tumor and pathological morphology using HE slides of lung tumor to determine the correlation between those variables. The tumor depth from the lung surface will be also collected to clarify the maximum depth to which the ultrasound can visualize.

SUMMARY:
The ex-vivo lung will be evaluated by XLTF-UC180 for localization of the tumor. The ultrasound probe will be put on the lung surface in several different directions to obtain the cross section with maximum diameter. The ultrasound image with size measurement of the tumor will be recorded using an ultrasound scanner (EU-Y0008, OLYMPUS MEDICALSYSTEMS CORP., Tokyo, Japan). Next, the bronchial stump of the specimen will be opened and a small sized endotracheal tube will be inserted to inflate and deflate the lung. After inflation of the lung, the tumor will be evaluated by XLTF-UC180 to see the difference in ultrasound images between deflated and inflated lung. After ultrasound evaluation, the specimen will be delivered directly to the pathology laboratory and the actual tumor size and histological diagnosis will be determined. In addition, we will evaluate the differences between US image and pathological morphology using HE slides of lung tumor. We will work together with the surgical team to confirm sign off of specimens.

DETAILED DESCRIPTION:
This is a single center clinical trial. Forty patients (sufficient for an initial evaluation) scheduled for a lobectomy or an anatomical segmental resection for malignant lung tumors will be enrolled in the study. After lung resection, the lung will be placed on a surgical table in a similar position to the in-vivo situation in the Image Guided Therapeutic operating room (GTx-OR) within Toronto General Hospital. The lung will be evaluated by XLTF-UC180 for localization of the tumor. The ultrasound probe will be put on the lung surface in several different directions to obtain the cross section with maximum diameter. The ultrasound image with size measurement of the tumor will be recorded using an ultrasound scanner (EU-Y0008, OLYMPUS MEDICALSYSTEMS CORP., Tokyo, Japan). Next, the bronchial stump of the specimen will be opened and a small sized endotracheal tube will be inserted to inflate and deflate the lung. After inflation of the lung, the tumor will be evaluated by XLTF-UC180 to see the difference in ultrasound images between deflated and inflated lung. After ultrasound evaluation, the specimen will be delivered directory to the pathology laboratory and the actual tumor size and histological diagnosis will be determined. In addition, we will evaluate the differences between US image and pathological morphology using Hemotoxylin and Eosin (HE) slides of lung tumor. We will work together with the surgical team to confirm sign off of specimens.

ELIGIBILITY:
Inclusion Criteria:

* Any patients scheduled for lobectomy of anatomical segmental resection for malignant lung tumors.
* 18 Years of age and older

Exclusion Criteria:

* Any patients with inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patients scheduled for lobectomy of anatomical segmental resection for malignant lung tumors.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2015-01; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Comparison of XLTF-UC180 Nodule Measurement with pathological morphology | 2 Years
  The primary objective of this study is to demonstrate the feasibility of thoracoscopic ultrasound for localization of pulmonary nodules in ex-vivo human lungs. We will evaluate the resected specimen using the XLTF-UC180 in the GTx-OR to determine the localization rate of the targets. Ultrasound measurement and images will be compared to the actual size of the tumor and pathological morphology using HE slides of lung tumor to determine the correlation between those variables. The tumor depth from the lung surface will be also collected to clarify the maximum depth to which the ultrasound can visualize

CONTACTS AND LOCATIONS:
Overall Officials: Kazuhiro Yasufuku, MD, PhD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Through Publication